CLINICAL TRIAL: NCT00546299
Title: Ambulatory Gas Usage in Patients With COPD and Exertional Hypoxemia
Brief Title: Gas Usage for Those With COPD Who Experience Low Oxygen Levels During Activities Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Collaborators: University of Toronto (Other); McMaster University (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8-42361
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2007-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Ambulatory oxygen therapy; COPD; exertional hypoxemia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oxygen — cylinder and concentrator, dosage to maintain SpO2 above 92%, used during exertion

SUMMARY:
Several studies have described the use of supplemental oxygen during exertion or activities of daily living (ambulatory oxygen) in study populations that have different characteristics. This report, based on specialized randomized controlled trials, characterizes ambulatory gas usage among patients with COPD who experience low oxygen levels during activities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* dyspnea limiting daily activities
* desaturation less than or equal to 88% for 2 continuous minutes during a room air six-minute walk test

Exclusion Criteria:

* less than or equal to 18 years old
* those who met criteria for mortality reduction with long-term oxygen
* those who received oxygen for palliative care or isolated nocturnal hypoxemia
* those unable to complete the questionnaires or provide informed consent

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-02; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
gas usage | 2

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, MD, Study Director — Respiratory Rehabilitation, West Park Healthcare Centre